CLINICAL TRIAL: NCT06882980
Title: Comparison of Ciprofol and Propofol Under IoC1 and IoC2 Monitoring for Adenotonsillectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy chief physician Investigator Affiliation Maternal and Child Health Hospital of Hubei Province, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MCHH_008
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Adenotonsillectomy; Propofol; Ciprofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol group (Experimental): Ciprofol group patients will be given ciprofol during anesthesia induction and maintenance
  Interventions: Other: Ciprofol group
- Propofol group (Active Comparator): Propofol group patients will be given propofol during anesthesia induction and maintenance
  Interventions: Other: Propofol group

INTERVENTIONS:
Other: Ciprofol group — In the Ciprofol group,children were given Ciprofol 0.6-0.8 mg/kg during anesthesia induction,and ciprofol 1.2-2 mg·kg-¹·h-¹for anesthesia maintenance.Throughout the entire process, we continuously monitor vital signs and IoC1/IoC2.
  Arms: Ciprofol group
Other: Propofol group — In the Propofol group,children were given Propofol 2.5-3.5 mg/kg during anesthesia induction,and propofol 6-10 mg·kg-¹·h-¹for anesthesia maintenance.Throughout the entire process, we continuously monitor vital signs and IoC1/IoC2.
  Arms: Propofol group

SUMMARY:
The goal of this clinical trial is to compare the Ciprofol and Propofol Under IoC1 and IoC2 Monitoring for Adenotonsillectomy Participants will be randomly allocated to two groups: Ciprofol group (Group C) and Propofol group (Group P). For those in Group C: they will be given ciprofol during anesthesia induction and maintenance .For those in Group P: they will be pgiven ciprofol during anesthesia induction and maintenanc This study evaluates ciprofol versus propofol under IoC1/IoC2 guidance in pediatric T&A, providing evidence for ciprofol's efficacy and safety in pediatric anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II, age 3-11 years, weight 13-50 kg.

Endoscopic T&A or adenoidectomy.

Exclusion Criteria:

* Recent upper respiratory infection.

Difficult airway, organ dysfunction, developmental/psychiatric disorders.

Drug allergies.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2025-11-22 (Estimated)

PRIMARY OUTCOMES:
Induction Compliance checklist(ICC) | during the time of anesthesia induction ,1 minute-10 minutes
  Induction Compliance checklist(ICC) will be recorded during the time of anesthesia induction.defined as a score out of 10.A score of 0 indicates perfect cooperation
The time to loss of consciousness during anesthesia induction | after the injection of anesthetic ,1second-5miutes
  The time to loss of consciousness during anesthesia induction will be recorded after the injection of anesthetic
sedation/consciousness (IoC1) | intraoperative period,10 minutes-1 hours
  sedation/consciousness (IoC1) will be recorded at 2 time points,including the time of intubation(T2) and mouth gag placement(T3)
analgesia/pain-stress (IoC2) | intraoperative period,10 minutes-1 hours
  analgesia/pain-stress (IoC2) will be recorded at 2 time points,including the time of intubation(T2) and mouth gag placement(T3)

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | intraoperative period,3 minutes-1 hour
  MAP will be monitored and recorded at 4 time points, including T1 (baseline), T2 (intubation), T3 (mouth gag placement), T4 (extubation)
Heart rate (HR) | intraoperative period,3 minutes-1 hour
  HR will be monitored and recorded at 4 time points, including T1 (baseline), T2 (intubation), T3 (mouth gag placement), T4 (extubation)
Recovery time | Postoperative 1 minutes to 1.5hours
  Time to fully awake. defined as by a modified Aldrete score which will be recorded with a recovery index of 9 to 26. The higher score means more awake.
Dosage of anesthetic | Intraoperative period, 20 minutes - 1.5 hours
  The total amount of sedative and analgesic drugs will be recorded.
anesthetist satisfaction | Postoperative 30 minutes
  Record the satisfaction of the anesthetist with the Ciprofol or Propofol ,defined as a score out of100.The higher score means more satisfaction
Adverse events | the procedure and Postoperative 24 hours
  The adverse events will be monitored and recorded during the operation and post-operation. AE will include:hypotension, bradycardia, respiratory depression, airway spasm, nausea, and vomiting
Pediatric Anesthesia Emergence Delirium (PAED) Scale | Postoperative 1 minute-1hour
  The Pediatric Anesthesia Emergence Delirium (PAED) Scale is a behavioral observation tool used to assess whether emergence delirium occurs in children after anesthesia. The total score ranges from 0 to 20.and a score of 10 or above is diagnostic of emergence delirium.A higher score indicates a greater tendency toward emergence delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes